CLINICAL TRIAL: NCT02296931
Title: Laboratory and Pilot Clinical Assessment of the Accuracy, Usability, and Function of a Low-cost, Low-power Syringe Pump in Administering Magnesium Sulfate to Pre-eclamptic Women in a Low-resource Hospital
Brief Title: Assessment of a Syringe Pump to Pre-eclamptic Women in a Low-resource Hospital
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Principal Investigator, Rebecca Richards-Kortum, Stanley C. Moore Professor, Bioengineering, William Marsh Rice University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-081F
Record Dates: First submitted 2014-11-18; First posted 2014-11-21 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Sodium Chloride; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Adults (Active Comparator): Phase 1 will be an initial validation of the clinical performance of the device delivering only standard IV saline to 10 stable women.
  Interventions: Other: Saline
- Pre-eclamptic pregnant women (Experimental): In Phase 2, the device will deliver MgSO4 to up to 40 women presenting with symptoms of pre-eclampsia.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Other: Saline — Standard IV Saline Fluids
  Arms: Healthy Adults
Drug: Magnesium Sulfate — The standard drug used to prevent and treat convulsions for women with pre-eclampsia and eclampsia is magnesium sulfate (MgSO4)
  Other Names: MgSO4
  Arms: Pre-eclamptic pregnant women

SUMMARY:
Pre-eclampsia and eclampsia cause 50,000 deaths annually. While MgSO4 is a widely accepted and relatively inexpensive treatment for these conditions, barriers to delivery via IV injection in low-resource settings pose a large obstacle to reductions in mortality. AutoSyP is a low-cost, low-powered automatic syringe pump that could overcome this barrier to the delivery of MgSO4. We propose to conduct a pilot clinical evaluation of its ability to deliver MgSO4 to women with pre-eclampsia or eclampsia in Malawi.

AutoSyP will be the subject of a 2 phase pilot clinical community trial in Malawi. Prior to the start of the study, all nurses will receive a 4-hour training on AutoSyP use to ensure proper procedures are followed. Phase 1 will be an initial validation of the clinical performance of the device delivering only standard IV saline to 10 stable women. The study will continue to Phase 2 where, the device will deliver MgSO4 to up to 40 women presenting with symptoms of pre-eclampsia.

1. Prior to the start of the study, all nurses will receive a 4-hour training on AutoSyP use.
2. Eligible and willing participants will provide informed consent. Then, baseline demographic and relevant medical history information will be collected.
3. In Phase 1, subjects will receive IV saline fluids by the Nurse. In Phase 2, the Nurse will provide loading dose of MgSO4 with the AutoSyP and research staff will monitor and record device performance and treatment specifications.
4. Subsequent maintenance doses of saline or MgSO4 will be administered and observations monitored and recorded for up to 24 hours as clinically indicated.

Others may benefit from this study in the future as AutoSyP is a new delivery system is needed to break down the barriers to IV delivery of MgSO4 in low-resource settings. The results of this study will be made available to the Ministry of Health, NHSRC, COMREC, the College of Medicine Library, the Department of Paediatrics, and other partners working in neonatal and child health. Findings will be published in academic journals and conference proceedings in an effort to disseminate results to potential end-users. The research findings of this study will be critical in the evaluation of future interventions.

DETAILED DESCRIPTION:
The study will recruit patients from two clinical sites (Kamuzu Central Hospital in Lilongwe, Malawi and Queen Elizabeth Central Hospital in Blantyre, Malawi) through their healthcare providers. Malawi represents an ideal location to conduct such a study as there are approximately 17,000 cases of pre-eclampsia annually. The study will include up to 40 women presenting with symptoms of pre-eclampsia.

The study will include pregnant women diagnosed with pre-eclampsia deemed to benefit from treatment with MgSO4 by healthcare providers at our participating clinical sites. Women who are eclamptic or seizing at the time of enrollment or have received MgSO4 therapy within the preceding 24 hours prior to study enrollment will be ineligible.

We will conduct an interventional study of the use of AutoSyP to deliver MgSO4 in two clinical setting in Malawi; Queen Elizabeth Central Hospital and Kamuzu Central Hospital. The study will be open and non-blinded due to ethical considerations that would arise from the denial of the experimental treatment to participants when there is no alternative form of IV MgSO4 delivery available.

All eligible and consenting women will be assigned to have treatment with AutoSyP if an AutoSyP device is available. If an AutoSyP device is not available, the participant will receive treatment for pre-eclampsia according to the standard of care at the hospital.

Pilot Clinical Evaluation Training

1. Prior to the start of the study, all nurses will receive a 4-hour training on AutoSyP use.
2. All trained nurses will receive an identification number that will be used for recordkeeping throughout the study.

Selection of Participants

1. Participants will be identified using the eligibility criteria stipulated above.
2. Willing participants will provide informed consent to participate in the study.
3. A participant identification number will be assigned. This number will be used for identification purposes throughout the study.
4. Baseline demographic and relevant medical history information will be collected.

Treatment

1. Nurse will provide loading dose with the AutoSyP. A trained Rice research assistant will observe all procedures and will correct any errors made by the nurse or answer any questions from the nurse.
2. The Rice research assistant will monitor the performance of the AutoSyP, watching for any device malfunctions and notify the nurse if any are observed. The Rice research assistant will help the nurse to correct the device malfunction and treatment will continue; otherwise, an alternative AutoSyP device will be used to continue treatment. The research assistant will also use a timer to record the duration of the dose.
3. The research assistant will record the following information:

   1. MgSO4 concentration used and syringe size
   2. Duration of administration
   3. Initial device set-up errors/questions by the nurse (e.g., user cannot operate device, user must ask for help)
   4. Observed malfunctions of AutoSyP
   5. Identification number of the nurse operating AutoSyP
   6. Identification number of the device
4. Nurse provides maintenance doses with AutoSyP after the loading dose is complete.
5. Rice research assistant repeats tasks 2-3 with reference to the maintenance dose.
6. Nurse continues to provide maintenance doses for up to 24 hours as necessary.
7. Rice research assistant repeats tasks 2-3 for each maintenance dose.
8. Treatment will be discontinued when clinically indicted.
9. Rice research assistant records the total number of doses provided and the clinical outcome of the patient.

ELIGIBILITY:
Phase 1: Healthy Volunteers

Inclusion Criteria:

* 18 years of age or older
* Provide informed consent
* Agree to comply with study procedures
* Deemed medically stable by their healthcare provider, including normal range blood pressure.
* Have been clinically identified to be able to receive standard IV saline fluid

Exclusion Criteria:

* Women with a history of heart disease of cardiac complications.
* Women with a history of complications with an IV.

Phase 2: Pre-eclamptic Women

Inclusion Criteria:

* 18 years of age or older
* Provide informed consent
* Agree to comply with study procedures
* Have systolic blood pressure P140mm Hg or a diastolic blood pressure P100mm Hg and proteinuria P1+.
* Be pregnant or are <24 hours postpartum.
* Diagnosed with pre-eclampsia and deemed to benefit from treatment with MGSO4 by healthcare providers

Exclusion Criteria:

* Have systolic blood pressure P140mm Hg or a diastolic blood pressure P100mm Hg and proteinuria P1+.
* Be pregnant or are <24 hours postpartum.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Kortum, PhD, Principal Investigator — William Marsh Rice University
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

REFERENCES:
- [Background] Duley L, Gulmezoglu AM, Henderson-Smart DJ, Chou D. Magnesium sulphate and other anticonvulsants for women with pre-eclampsia. Cochrane Database Syst Rev. 2010 Nov 10;2010(11):CD000025. doi: 10.1002/14651858.CD000025.pub2. PMID 21069663
- [Background] Connor SB, Quill TJ, Jacobs JR. Accuracy of drug infusion pumps under computer control. IEEE Trans Biomed Eng. 1992 Sep;39(9):980-2. doi: 10.1109/10.256432. PMID 1473827
- [Derived] Skerrett E, Kommwa E, Maynard K, Juarez A, Mataya R, Richards-Kortum R, Oden ZM. Evaluation of a low-cost, low-power syringe pump to deliver magnesium sulfate intravenously to pre-eclamptic women in a Malawian referral hospital. BMC Pregnancy Childbirth. 2017 Jun 19;17(1):191. doi: 10.1186/s12884-017-1382-9. PMID 28629437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Adults | Pre-eclamptic Pregnant Women
Started | 10 | 24
Completed | 10 | 22
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Adults | Pre-eclamptic Pregnant Women | Total
Number analyzed (Participants) | 10 | 22 | 32
Age, Continuous [Median (Full Range); unit: years] | 28 [23 to 50] | 26 [19 to 37] | 27 [19 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 10 | 22 | 32

OUTCOME MEASURES:

1. Primary Outcome: Error in the Total Volume Dispensed and Flow Rate
Description: This is the error value for the volume dispensed by the AutoSyp device relative to the volume intended to be dispensed. Preeclamptic subjects received an initial loading dose followed by a maintenance dose. The loading dose had a flow rate of 60 mL/hr and delivered 20 mL in a single 20 mL syringe. The maintenance dose was 5 mL/hr and dispensed 120 mL total through two 60 mL syringes. The healthy subjects experienced variable flow rates and dispensed volumes, so they do not have the same variables as the pre-eclamptic pregnant women in the outcome data tables below. Because of these differences in dosing the two arms of the study, healthy women and preeclamptic women have different outcome measure data.
Time Frame: 1 day visit
Measure: Mean (Full Range); unit: percentage of error
Arm/Group | Healthy Adults | Pre-eclamptic Pregnant Women
Number analyzed (Participants) | 10 | 22
percentage of error
  Total Volume Dispensed-Loading Dose | NA [NA to NA] — Healthy adults experienced variable dispensed volumes in contrast to the fixed volumes dispensed for the pre-eclamptic arm. This category is only for the error experienced by the pre-eclamptic arm regarding their fixed loading dose volume of 20mL | -1.48 [-2.58 to -0.58]
  Flow Rate-Loading Dose | NA [NA to NA] — Healthy adults experienced variable flow rates in contrast to the fixed flow rates of the pre-eclamptic arm. This category is only for the error experienced by the pre-eclamptic arm regarding their loading dose flow rate of 60mL/hr. | -1.75 [-2.53 to -1.47]
  Total Volume Dispensed-Maintenance Dose | NA [NA to NA] — Healthy adults had variable dispensed volumes in contrast to the fixed volumes dispensed for the pre-eclamptic arm. This category is for the error experienced by the pre-eclamptic arm regarding their maintenance dose dispensed volume of 120mL . | -1.13 [-2.28 to -0.41]
  Flow Rate-Maintenance Dose | NA [NA to NA] — Healthy adults experienced variable flow rates in contrast to the fixed flow rates for the pre-eclamptic arm. This category is only for the error experienced by the pre-eclamptic arm regarding their maintenance dose flow rate of 5mL/hr. | -1.11 [-2.09 to -0.76]
  Flow Rate-Variable | -0.21 [-2.90 to 4.95] | NA [NA to NA] — Healthy adult women experienced variable flow rates in contrast to the fixed flow rates for the pre-eclamptic arm. This category is only for the variable flow rate error experienced by the health adult arm.
  Total Volume Dispensed-Variable | -1.07 [-3.65 to 2.60] | NA [NA to NA] — Healthy adult women experienced variable dispensed volumes in contrast to the fixed volumes dispensed for the pre-eclamptic arm. This category is only for the error in total volume dispensed experienced by the healthy adult arm.

ADVERSE EVENTS:
Arm/Group | Healthy Adults | Pre-eclamptic Pregnant Women
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/24
Other Adverse Events (participants affected / at risk) | 0/10 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No